### Title:

# Role of Triceps Kinesiology Taping on Elbow Flexion Tightness in Extended Erb's Palsy Infants

NCT: not yet assigned

Document Date: 05/06/2018

# FACULTY OF PHYSICAL THERAPY APPLICATION FOR ETHICAL REVIEW

#### NOTES:

- Answers to questions must be entered in the space provided.
- An electronic version of the completed form should be submitted to the Research Ethics

  Officer, at the following email address: <a href="mailto:...ethical@pt.cu.edu.eg.....">...ethical@pt.cu.edu.eg.....</a>. Please **do not** submit paper copies.
- ➤ If you have any queries about the form, please address them to the Research Ethics Team .

## FACULTY OF PHYSICAL THERAPY APPLICATION FOR ETHICAL REVIEW

OFFICE USE ONLY:
Application No:
Date Received:

| 1. | TITL | .E ( | )F | PR( | OP | OSAL |
|----|------|------|----|-----|----|------|
|----|------|------|----|-----|----|------|

ROLE OF TRICEPS KINESIOLOGY TAPING ON ELBOW FLEXION TIGHTNESS IN EXTENDED ERB'S PALSY INFANTS

| . THIS PROPOSAL IS: | | | |
|---|---|---|---|
| Physical Therapy Staff Research P | roposal 🔲 | | |
| Physical Therapy Postgraduate Research (PGR) tudent Proposal √ | | | |
| | Master <sup>□</sup> | Doctoral $\sqrt{}$ | Other |
| Other Please specify): | | | |

#### 3. INVESTIGATORS

# a) PLEASE GIVE DETAILS OF Student (FOR PGR STUDENT PROPOSAL) or first author for staff Research Proposal

| Name: Title / first name / family name | Radwa Said Shahat Ahmed |
|---|---|
| Highest qualification & position held: | MSc. Of Pediatric Physical Therapy, Assistant Lecturer at MTI University |
| Department/ Faculty/ University Telephone: | Pediatrics/Physical Therapy/MTI university |
| Email address: | +2 01004008503 |
| | radwasaid@live.com |

## a) PLEASE GIVE DETAILS OF ANY CO-SUPERVISORS OR CO-INVESTIGATORS (FOR PGR STUDENT PROPOSAL) or co- first author for staff Research Proposal b)

| Name: Title / first name / family name | Prof. Emam Hassan Elnegmy |
|---|---|
| Highest qualification & position held: | Professor |
| Department/ Faculty/ University Telephone: | Pediatrics/Physical Therapy/ Cairo University |
| Email address: | |
| | Emamhassan20@yahoo.com |
| Name: Title / first name / family name | Prof. Gehan Mosaad Abd ElMaksoud |
| Highest qualification & position held: | Professor |
| Department/ Faculty/ University Telephone: | Pediatrics/Physical Therapy/ Cairo University |
| Email address: | |
| | Gehanmosaad@gmail.com |

| Name: Title / first name / family name | Prof. Amena Mohamed Hindawy |
|---|---|
| Highest qualification & position held: | Professor |
| Department/ Faculty/ University Telephone: Email address: | Pediatrics/Medicine/ Cairo University |

#### 4. SUMMARY OF PROPOSAL

To determine the role of using Kinesiology tape on the prevention of elbow flexion tightness in infants with extended Erb's palsy.

#### **PURPOSE:**

To determine the role of using Kinesiology tape on the prevention of elbow flexion tightness in infants with extended Erb's palsy.

#### **BACKGROUND:**

Neglecting or even delay in BPBP management, may result in substantial and chronic impairment. Physiotherapy, microsurgical nerve reconstruction, secondary joint corrections, and muscle transpositions are employed to help the child maximize function in the affected upper extremity. Kinesiology taping can have an effect on muscle performance and support joint by improving proprioception, normalizing muscle tone, correct the inappropriate positions and stimulate skin receptors. The possible effect of KT on muscle strength has been investigated by numerous researchers that have theorized that KT facilitates an immediate increase in muscle strength by generating a concentric pull on the fascia.

#### **HYPOTHESES:**

There will be no role of Kinesiology tape on the prevention of elbow flexion tightness in infants with extended Erb's palsy.

#### **RESEARCH QUESTION:**

Is there a role of using Kinesiology tape in preventing elbow flexion tightness in infants with extended Erb's palsy?

#### 5. CONDUCT OF PROJECT

#### Please give a description of the research methodology that will be used

- 1. Toronto active motion scale will be used to determine functional strength of the Biceps and Triceps Brachii muscles.
- 2. The G-Pro application will be downloaded on the smartphone and used to measure the range of motion of elbow extension.
- 3. A computerised electromyographic apparatus (Neuroscreen plus 4 channel version 1.59 produced by TOENNIES, 97204 Hochberg, Germany) will be used to measure the percentages of degeneration of the Biceps and Triceps Brachii muscles using surface electrodes.
- 4. Kinesiology Taping will be used as a facilitator to the Triceps muscle (as treatment along a traditional Physical Therapy treatment program). One I-shaped tape will be taped over the triceps muscle.

#### 6. PARTICIPANTS AS THE SUBJECTS OF THE RESEARCH

Describe the number of participants and important characteristics (such as age, gender, intellectual ability etc.). Specify any inclusion/exclusion criteria to be used.

Thirty two infants of both genders will be recruited.

Ages range from 3-6 months of age.

They will be diagnosed with Obstetric Brachial Plexus palsy- Extended Erb's Palsy (C5-6-7)

#### 7. RECRUITMENT

Please state clearly how the participants will be identified, approached and recruited.

Note: Attach a copy of any poster(s), advertisement(s) or letter(s) to be used for recruitment.

- Patients will have unilateral extended brachial plexus injury involving cervical 5, 6 and 7 roots lesion.
- 2. They will have positive grasp reflex.
- 3. They will have asymmetrical Moro reflex.
- 4. They will show evidence of degeneration of both the Triceps and Biceps Brachii muscles.

Patients will be selected, evaluated and treated at the outpatient clinics of the Faculties of Physical Therapy of both Cairo University and Modern University for Information and Technology.

#### 8. CONSENT

Describe the process that the investigator(s) will be using to obtain valid consent. If consent is not to be obtained explain why. If the participants are minors or for other reasons are not competent to consent, describe the proposed alternate source of consent, including any permission / information letter to be provided to the person(s) providing the consent.

| I am<br>M.Sc. | freely and voluntarily consent to participate in a research program under the direction of |
|---|---|
| | ugh description of the procedure has been explained and I understand that I may withdraw my<br>t and discontinue participation in this research at any time without prejudice to me.<br>Participant |
| Noto: | Attach a copy of the Consent Form, Participant Information Sheet (if applicable). |
| wote: | Attach a copy of the Consent Form, Participant Information Sheet (ii applicable). |
| DARTIC | IPANT WITHDRAWAL |
| | ibe how the participants will be informed of their right to withdraw from the project. |
| a) Desci | the now the participants will be informed of their right to withdraw from the project. |
| They ca | an withdraw at anytime without prejudice to them as mention in signed consent. |
| THEY Co | an withdraw at anytime without prejudice to them as mention in signed consent. |
| n) Expla | in any consequences for the participant of withdrawing from the study and indicate what |
| will | be done with the participant's data if they withdraw. |
| No cons | sequences will take place. They have the utmost freedom. |
| . 40 0011 | bequestions will take place. They have the difficult freedom. |

#### 9. CONFIDENTIALITY

| a) | Will all participants be anonymous? | Yes $\sqrt{\ }$ | No 🖳 | |
|----|-------------------------------------------|-----------------|------|---|
| b) | Will all data be treated as confidential? | Yes $\sqrt{\ }$ | No 💾 | Ш |

Note: Participants' identity/data will be confidential if an assigned ID code or number is used, but it will not be anonymous. Anonymous data cannot be traced back to an individual participant.

#### 10. SIGNIFICANCE/BENEFITS

Outline the potential significance and/or benefits of the research

Delay in the treatment of extended Erb's palsy may result in substantial and chronic impairment due to many causes. One of the causes is the imbalance between the recovery of elbow lexors and elbow extensors where the latter will be delayed. This study will determine if a debilitating tightness and contracture (elbow flexion) can be prevented using the kinesiology tape in infants with Extended Erb's Palsy.

#### **11. RISKS**

Outline any potential risks to **INDIVIDUALS**, including research staff, research participants, other individuals not involved in the research and the measures that will be taken to minimise any risks and the procedures to be adopted in the event of mishap

Risk of Infection: minimizing the risk through adequate sterilization of the treated areas during evaluation and treatment.

#### 12. DECLARATION BY APPLICANTS

I submit this application on the basis that the information it contains is confidential and will be used by the Faculty of Physical Therapy for the purposes of ethical review and monitoring of the research project described herein, and to satisfy reporting requirements to regulatory bodies. The information will not be used for any other purpose without my prior consent.

#### I declare that:

- The information in this form together with any accompanying information is complete and correct to the best of my knowledge and belief and I take full responsibility for it.
- I will report any changes affecting the ethical aspects of the project to the Faculty of Physical Therapy Research Ethics Officer.
- I will report any adverse or unforeseen events which occur to the relevant Ethics Committee via the Faculty of Physical Therapy Research Ethics Officer.

| Name of Principal investigator/project supervisor: | Radwa Said Shahat Ahmed |
|---|---|
| | Prof. Emam Hassan ElNegmy |
| Date: | 6 <sup>th</sup> of May, 2018 |